CLINICAL TRIAL: NCT04963868
Title: Timing of Transmural Stent Removal in Necrotizing Pancreatitis Undergoing Endoscopic Transmural Necrosectomy: A Randomized Controlled Study
Brief Title: Timing of Transmural Stent Removal in Necrotizing Pancreatitis
Acronym: TTSRNP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The First Affiliated Hospital of Nanchang University (Other)
Responsible Party: Principal Investigator, Lingyu Luo, Physician-in-charge, The First Affiliated Hospital of Nanchang University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FAH of NCU
Record Dates: First submitted 2021-06-21; First posted 2021-07-15 (Actual); Last update posted 2021-07-15 (Actual); Status verified 2021-07

CONDITIONS: Acute Pancreatitis; Necrotizing Pancreatitis; Walled-Off Necrosis
Keywords: Necrotizing pancreatitis; Endoscopic transmural necrosectomy; Lumen-apposing metal stent
MeSH Terms: conditions — Pancreatitis; Pancreatitis, Acute Necrotizing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The novel strategy group (Experimental): The stents were removed during the last necrosectomy when the endpoint of necrosectomy was achieved
  Interventions: Procedure: Stent removed by the novel strategy
- The conventional strategy group (Active Comparator): The stent was removed after the last necrosectomy when clinical symptoms were relieved and fluid was nearly completely resolved confirmed by CT image
  Interventions: Procedure: Stent removed by the conventional strategy

INTERVENTIONS:
Procedure: Stent removed by the novel strategy — The stent was removed during the last necrosectomy when the endpoint of necrosectomy was achieved；
  Arms: The novel strategy group
Procedure: Stent removed by the conventional strategy — The stent was removed after the last necrosectomy when clinical symptoms were relieved and fluid was nearly completely resolved confirmed by CT image.
  Arms: The conventional strategy group

SUMMARY:
Although metal stents have been widely used in the endoscopic step-up approach for necrotizing pancreatitis, the exact timing of transmural stent removal has not been well studied. In this prospective, open-label, randomized controlled study, we recruited and enrolled consecutive patients with necrotizing pancreatitis undergoing endoscopic transmural necrosectomy. Eligible participants were randomly assigned to case group (a novel strategy in which the stents were removed during the last necrosectomy when the necrosectomy endpoint was achieved) and control group (the conventional strategy in which the stents were removed after the last necrosectomy when clinical symptoms were relieved and fluid was nearly completely resolved confirmed by imaging). The primary endpoint was the incidence of composite complications within three months of enrollment.

DETAILED DESCRIPTION:
Over the last decade, approaches to managing necrotizing pancreatitis have evolved from open surgery to a minimally invasive approach due to the efficacy and lower morbidity and mortality rates of the latter technique. As one of minimally invasive approaches, endoscopic step-up approach, with transmural drainage whenever feasible and subsequent necrosectomy as required, was first described in 1996 and has evolved to first-line therapy for symptomatic necrotizing pancreatitis. However,The exact timing of transmural stent removal has not been well studied. The conventional strategy for stent removal in the published guidelines has been that patients should undergo follow-up imaging and stent removal at 4-8 weeks if walled-off necrosis has resolved. Here, we introduced a novel strategy in which the stents were removed during the last necrosectomy when the endpoint of endoscopic transmural necrosectomy was achieved, that was, the necrotic tissue was nearly completely removed, and the pink granulation tissue lining the wall was uncovered. Compared to the conventional strategy, the novel strategy avoided one endoscopy procedure. The present study is the first prospective, open-label, randomized controlled study to investigate the efficacy and safety of the novel strategy. We recruited and enrolled consecutive patients with necrotizing pancreatitis undergoing endoscopic transmural necrosectomy. Eligible participants were randomly assigned to case group (a novel strategy in which the stents were removed during the last necrosectomy when the necrosectomy endpoint was achieved) and control group (the conventional strategy in which the stents were removed after the last necrosectomy when clinical symptoms were relieved and fluid was nearly completely resolved confirmed by imaging). The primary endpoint was the incidence of composite complications within three months of enrollment.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with necrotizing pancreatitis according to the 2012 Atlanta classification criteria;
2. Patients aged between 18 and 65 years;
3. Patients who signed the informed consent;

Exclusion Criteria:

1. Patients without transmural stent placement;
2. Patients with transmural plastic stent not metal stent placement before enrollment;
3. Patients who underwent endoscopic transmural necrosectomy in other hospitals before admission;
4. Patients complicated with chronic pancreatitis;
5. Patients complicated with pancreatic tumor;
6. Pregnant or lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Estimated)
Dates: Start 2022-01-01 (Estimated); Primary Completion 2024-06-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
The incidence of composite complications | 3 months
  The composite complications included new-onset organ failure or systemic complications、new-onset infectious pancreatic necrosis、abdominal or gastrointestinal bleeding, intestinal fistula, stent occlusion and stent migration.

SECONDARY OUTCOMES:
The incidence of technical success | 3 months
  Technical success was defined by stent removed successfully.
The incidence of clinical success | 3 months
  Clinical success was defined as nearly completely resolution or <2 cm of collection assessed by image at the three-month follow-up without additional open surgery or death.
The number of endoscopic transmural necrosectomy sessions | 3 months
  Total sessions of patients undergoing endoscopic transmural necrosectomy.
The number of additional endoscopic transmural necrosectomy sessions after stent removal | 3 months
  Additional sessions of patients undergoing endoscopic transmural necrosectomy. after stent removal.
Length of stent placement | 3 months
  The duration time from stent placement to stent removal.
The incidence of open surgery | 3 months
  The incidence of patients needing open surgery after minimally invasive treatment.
All-cause mortality | 3 months
  The mortality whatever the cause is.
Length of hospital stay | 3 months
  The length of hospital stay due to necrotizing pancreatitis.
The incidence of readmission | 12 months
  The incidence of readmission after index discharge due to pancreatitis related problems.
The hospital cost | 3 months
  The hospital cost during hospitalization.

CONTACTS AND LOCATIONS:
Overall Officials: Yin Zhu, PhD, Principal Investigator — The First Affiliated Hospital of Nanchang University
Locations (1):
- The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi, China